CLINICAL TRIAL: NCT02053857
Title: A Randomized, Double-blind Pilot Study of Polyunsaturated Fatty Acid-optimized Ready-to-use Therapeutic Food, Compared to Standard RUTF, in the Therapy of Severe Acute Malnutrition
Brief Title: Pilot Study of PUFA-optimized RUTF for Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUFA-RUTF Pilot
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Kwashiorkor; Marasmus
Keywords: severe acute malnutrition; polyunsaturated fatty acids; ready-to-use therapeutic food
MeSH Terms: conditions — Kwashiorkor; Protein-Energy Malnutrition; Severe Acute Malnutrition | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RUTF (Active Comparator): Standard RUTF at a dose of 175 kcal/kg/d
  Interventions: Dietary Supplement: RUTF; Drug: Amoxicillin
- RUTF-P (Experimental): RUTF fortified with polyunsaturated fatty acids (PUFA) at a dose of 175 kcal/kg/d
  Interventions: Dietary Supplement: RUTF-P; Drug: Amoxicillin

INTERVENTIONS:
Dietary Supplement: RUTF
  Other Names: ready-to-use therapeutic food
  Arms: RUTF
Dietary Supplement: RUTF-P
  Arms: RUTF-P
Drug: Amoxicillin

SUMMARY:
To test whether a ready-to-use therapeutic food (RUTF) enriched with polyunsaturated fatty acids (RUTF-P) is as effective for the treatment of severe acute malnutrition (SAM) as standard RUTF.

DETAILED DESCRIPTION:
Since 2007, RUTF has been the recommended treatment for SAM. RUTF is not conducive to the growth of bacteria because of the low moisture content, does not require cooking, and has led to greater recovery rates than liquid milk formulations in direct comparisons. One expected benefit of the RUTF-P is improved outcomes due to the higher levels of essential fatty acids.

The essential fatty acid profile (i.e., the level of omega-3 and omega-6 fatty acids) of RUTF-P may have important implications for cognitive development of children, especially infants, with SAM who consume these foods as their sole dietary source for several weeks. In particular, an excess of omega-6 fatty acids (from sources such as peanut and corn oil) and a minimum of omega-3 fatty acids (from sources like flax) may fail to support optimal cognitive development and neural function.

In this prospective, double-blinded, randomized controlled clinical effectiveness trial, we will compare two RUTF products in the treatment of SAM to test the effects of the two different RUTF products on essential fatty acid status.

ELIGIBILITY:
Inclusion Criteria:

* kwashiorkor and/or marasmus
* 6-59 months of age
* lives in local area near enrollment site

Exclusion Criteria:

* recent (<4 months) therapeutic feeding for moderate or severe acute malnutrition
* chronic medical condition (eg, Down syndrome, other congenital syndrome, chronic heart disease) that may make feeding and growth difficult (not to include HIV or TB)
* caretaker refusal of 2 blood draws
* ineligibility for outpatient therapy (ie, severe illness or anorexia requiring inpatient therapy)
* caretaker expresses plans to move away from local area of clinic, making followup difficult

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
DHA Level | 4 weeks
  Blood plasma docosahexaenoic acid (DHA) levels
EPA Level | 4 weeks
  Blood plasma eicosapentaenoic acid (EPA) levels

SECONDARY OUTCOMES:
Recovery Rate | 12 weeks
  Proportion of children who recover from SAM
Linear Growth | 12 weeks
  Changes in length
Ponderal Growth | 12 weeks
  Changes in weight
Growth | 12 weeks
  Changes in mid-upper-arm circumference

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine; Kenneth Maleta, MBBS PhD, Principal Investigator — University of Malawi; Chrissie Thakwalakwa, Principal Investigator — University of Malawi
Locations (1):
- University of Malawi College of Medicine, Blantyre, Malawi